CLINICAL TRIAL: NCT03544996
Title: A Comparison of Injected Insulin Replacement Therapy With A Novel Transdermally Delivered Human Insulin Product
Brief Title: Transdermally Delivered Human Insulin Product
Status: Completed | Type: Observational
Sponsor: Transdermal Delivery Solutions Corp (Industry)
Responsible Party: Sponsor
Other Study IDs: TDS INS-001
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Hypoinsulinemia
Keywords: Insulin, needle-less, transdermal
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TD Insulin Pilot: Test of novel transdermal insulin (TD Insulin) formulations
  Interventions: Combination Product: TD Insulin

INTERVENTIONS:
Combination Product: TD Insulin — Human Insulin USP formulated in a solution capable of transdermal delivery.

SUMMARY:
An Early Feasibility Study of a device formulation to deliver human insulin across intact skin

DETAILED DESCRIPTION:
An attempt was made to formulate an insulin product that would complex human insulin in a stable anhydrous solution and when applied to the skin enable the uptake and release of insulin in a brittle T1D patient.

A series of formulations were produced at varing dose strengths and in conjunction with injected insulin products, applied and serum glucose measured to ascertain response and optimize a fomrula to be submitted for IND approval.

ELIGIBILITY:
Inclusion Criteria:

* Brittle T1D patient with poor insulin sensitivity requiring more than 3,000 IUs on insulin a day

Exclusion Criteria:

* High insulin sensitivity
* well managed serum glucose

Ages: 60 Years to 61 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Single patient, brittle T1D patient
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-02-04 (Actual); Study Completion 2018-02-04 (Actual)

PRIMARY OUTCOMES:
Insulin response | 8-24 hours
  Measurement of down modulation of serum glucose as measured by a standard blood glucose meter not otherwise attributable to injected insulin

CONTACTS AND LOCATIONS:
Overall Officials: William D Kirsh, D.O., Principal Investigator — Sentry Data Systems
Locations (1):
- Langford Research Institute, Palm Beach Gardens, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided